CLINICAL TRIAL: NCT05481515
Title: A Study Within a Trial to Determine the Effect of Skin Tone on the Diagnostic Accuracy of Pulse Oximeters
Brief Title: Exploring Pulse OXimeter Accuracy Across SKin Tones
Acronym: EXAKT
Status: Completed | Type: Observational
Sponsor: Intensive Care National Audit & Research Centre (Other)
Collaborators: Lewisham Council (Unknown); Centre Ethnic Health Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: EXAKT Sub-Study
Record Dates: First submitted 2022-07-22; First posted 2022-08-01 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Critical Illness; Hypoxemia
MeSH Terms: conditions — Critical Illness; Hypoxia | interventions — Oximetry; Spectrophotometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Critically ill adults: Adult patients admitted to an intensive care unit who require mechanical ventilation and supplemental oxygen
  Interventions: Device: Pulse oximetry; Device: Spectrophotometry

INTERVENTIONS:
Device: Pulse oximetry — Pulse oximeters will be evaluated against routine arterial blood gas measurements
Device: Spectrophotometry — Spectrophotometry will be used to measure skin tone

SUMMARY:
This study within a trial (SWAT) will be a sub-study of the UK-ROX trial (ISRCTN13384956), which is currently running in intensive care units across the UK. UK-ROX is large-scale randomised controlled trial evaluating conservative oxygen therapy (a target SpO2 of 88-92%) versus usual oxygen therapy in mechanically ventilated adult patients admitted to ICUs in the UK. The purpose of this observational sub-study is to compare pulse oximeter-derived peripheral oxygen saturation (SpO2) values to co-oximeter-derived arterial oxygen saturation (SaO2) measurements from arterial blood gas (ABG) samples, for a range of fingertip pulse oximeters in an ethnically diverse group of adult patients admitted to UK intensive care units (ICUs). Approximately 900 patients will be recruited over 12 month period from 24 sites to provide an anticipated 10,800 paired SpO2 and SaO2 measurements. Patient skin tone will be objectively measured using a handheld spectrophotometer. Data from the sub-study will be used to determine the accuracy of the tested pulse oximeters across a range of skin tones and arterial oxygenation levels.

DETAILED DESCRIPTION:
Research question: What is the diagnostic accuracy of different pulse oximeters at peripheral oxygen saturation levels (SpO2) relevant to their use by patients at home and how does this vary in people with darker skin pigmentation?

Primary objective: To compare pulse oximeter-derived SpO2 values to co-oximeter-derived arterial oxygen saturation (SaO2) measurements from arterial blood gas (ABG) samples, for a range of fingertip pulse oximeters in an ethnically diverse group of adult patients with a broad spectrum of skin tones admitted to UK intensive care units (ICUs).

Design: This study within a trial (SWAT) that will form an observational sub-study of the NIHR HTA funded UK-ROX trial (https://fundingawards.nihr.ac.uk/award/NIHR130508), which is currently running in ICUs across the UK. Twenty four ICUs enrolling patients into the UK-ROX trial trial will be randomly allocated two brands of pulse oximeter to evaluate. Over a period of 24 hours for each participant, SpO2 values from the test pulse oximeters will be compared to simultaneous SaO2 values from ABG samples analysed on a standard ICU ABG co-oximeter machine. Patient skin tone will be objectively measured using a handheld spectrophotometer. The difference between SpO2 and SaO2 will be compared across skin tones and across a range of arterial oxygenation levels.

Setting: The UK-ROX trial is large-scale, multi-centre, data-enabled, registry embedded randomised controlled trial (RCT) evaluating conservative oxygen therapy (a target SpO2 of 88-92%) versus usual oxygen therapy in mechanically ventilated adult patients admitted to ICUs in the United Kingdom.

Target population: 900 mechanically ventilated adults screened for enrolment into the UK-ROX trial.

Primary outcome: The accuracy of SpO2 measurement in the evaluated pulse oximeters, validated against co-oximeter-derived SaO2 ABG sample analysis.

ELIGIBILITY:
Inclusion Criteria are for those of the main UK-ROX trial:

* Adult (aged ≥18 years)
* Receiving invasive mechanical ventilation in the ICU following an unplanned ICU admission OR invasive mechanical ventilation started in the ICU (i.e. the patient was intubated in the ICU).
* Receiving supplemental oxygen (> 21% oxygen) at the time of enrolment

Exclusion Criteria are for those of the main UK-ROX trial:

• The clinician considers that one study treatment arm is either indicated or contraindicated.

In order in increase the number of patients eligible for this observational diagnostic accuracy study, we will have also received ethical approval to enrol mechanically ventilated adult patients who have been screened for, but not enrolled into, the UK-ROX trial. These may include patients who missed the 12 hour recruitment window for the main trial and patients in whom the clinical team decided that one study treatment arm is either indicated or contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to an ICU who require mechanical ventilation and supplemental oxygen.
Sampling Method: Non-Probability Sample
Enrollment: 903 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of SpO2 measurements | Over 24 hour observation window
  Accuracy of SpO2 measurement, validated against co-oximeter derived SaO2 arterial blood gas analysis (calculated as SpO2 minus paired SaO2)

SECONDARY OUTCOMES:
Detection of hypoxaemia | Over 24 hour observation window
  Diagnostic accuracy (area under the receiver operating characteristic curve and sensitivity and specificity at relevant cut-points) for SpO2 as a predictor of SaO2 ≤ 92%.
Detection of occult hypoxaemia | Over 24 hour observation window
  The presence of an SaO2 < 88% among participants with a paired SpO2 reading of >92%

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care National Audit and Research Centre, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
If requested, we aim to make the IPD data available to other investigators. This will include anonymised data related to the accuracy of the tested pulse oximeters.

REFERENCES:
- [Derived] Martin DS, Doidge JC, Gould D, Shahid T, Cowden A, Charles WN, Francis Johnson A, Garrett R, Mbema C, Olusanya O, Healy E, Rowan K, Mouncey P, Harrison DA; EXAKT Study Investigators. The impact of skin tone on performance of pulse oximeters used by NHS England COVID Oximetry @home scheme: measurement and diagnostic accuracy study. BMJ. 2026 Jan 14;392:e085535. doi: 10.1136/bmj-2025-085535. PMID 41534914